CLINICAL TRIAL: NCT06359210
Title: An Adaptive Physical Activity Maintenance Intervention
Brief Title: Sustaining Physical Activity After Cancer Exercise Sessions
Acronym: SPAACES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Heather Leach, Associate Professor, Colorado State University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4973; 4R33CA256656-03 (NIH)
Record Dates: First submitted 2024-03-20; First posted 2024-04-11 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Exercise Oncology; Physical Activity Behavior; Behavior Change Interventions
Keywords: exercise oncology; physical activity; behavior change; adaptive intervention; cancer survivors; physical activity maintenance; community partnerships
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: An adaptive design results in a final total of 4 possible subgroups, depending upon responder/non-responder status, and researchers plan to compare the proportion of participants achieving the minimum exercise guidelines for cancer survivors within the responders and incomplete responder subgroups. Admittedly however, it is not possible to fully elucidate the analyses the researchers will conduct, as researchers cannot predict the number of subgroups that participants will represent at the end of the trial (e.g., if there are no "incomplete responders" the design reduces to randomization to only two groups), nor the number of participants who will be in those subgroups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A- Complete Responder (No Intervention): Participant is randomized to the no further intervention group.
- Group B- Complete Responder (Experimental): Participant is randomized to receive monthly physical activity behavior change discussion sessions for 3-months (total of three sessions).
  Interventions: Behavioral: Responder Monthly Behavior Change Discussion Sessions
- Group C- Incomplete Responder (Experimental): Participant is randomized to receive monthly physical activity behavior change discussion sessions for 3-months (total of three sessions).
  Interventions: Behavioral: Incomplete Responder Monthly Behavior Change Discussion Sessions
- Group D- Incomplete Responder (Experimental): Participant is randomized to receive monthly physical activity behavior change discussion sessions for 3-months (total of three sessions) AND bi-weekly exercise sessions (total of six sessions).
  Interventions: Behavioral: Incomplete Responder Monthly Behavior Change Discussion Sessions + Bi-Weekly Exercise Sessions

INTERVENTIONS:
Behavioral: Responder Monthly Behavior Change Discussion Sessions — Monthly behavior change discussion sessions (3 total) for 12 weeks.
  Arms: Group B- Complete Responder
Behavioral: Incomplete Responder Monthly Behavior Change Discussion Sessions — Monthly behavior change discussion sessions (3 total) for 12 weeks.
  Arms: Group C- Incomplete Responder
Behavioral: Incomplete Responder Monthly Behavior Change Discussion Sessions + Bi-Weekly Exercise Sessions — Monthly behavior change discussion sessions (3 total) for 12 weeks and attend bi-weekly (every other week) exercise classes that mirror the exercises completed in their respective community-based exercise program.
  Arms: Group D- Incomplete Responder

SUMMARY:
The goal of this clinical trial is to develop and test an adaptive physical activity (PA) maintenance intervention for cancer survivors, after participating in a community-based exercise oncology program. The main questions it aims to answer are:

* Aim 1: Examine the feasibility and acceptability of the intervention among cancer survivors and community partners. The researchers will utilize quantitative surveys, focus groups, and semi-structured interviews to collect information about feasibility, implementation, adaptation, and sustainability.
* Aim 2: Examine the effects of the intervention among cancer survivors. The researchers will compare the proportion of participants achieving the exercise guidelines for cancer survivors six-months following completion of the initial exercise program.

Participants will participate in a community-based exercise oncology program and then return to three months of free living. Based on the PA measured at the three-month follow-up, participants will be categorized as a "Responder" or "Incomplete Responder", and then randomized to the PA maintenance intervention. Researchers will compare those that are classified as Responders (meeting exercise guidelines for cancer survivors) and Incomplete Responders (not meeting guidelines for cancer survivors) to see what level of intervention is needed to influence sustainable behavior change in this population.

DETAILED DESCRIPTION:
Structured leisure-time physical activity (PA) (i.e., aerobic and resistance exercise) is effective for improving multiple health outcomes related to a cancer diagnosis and cancer treatment and may reduce cancer-specific mortality by as much as 40%. Thus, if cancer survivors can achieve and maintain recommended exercise levels, the public health impact would be substantial.

Supervised exercise interventions that include theory-based behavior change strategies are effective for facilitating increases in moderate to vigorous, leisure-time PA among cancer survivors. However, few studies have focused on maintaining exercise or PA levels following completion of an intervention, and evidence regarding how exercise interventions for cancer survivors can be expanded to clinic or community practice is only now emerging. To achieve the physical, psychosocial, and survival benefits of exercise, survivors must be able to maintain PA long-term, and to support PA maintenance, a socio-ecological approach is necessary. Our approach is informed by theoretical frameworks including social cognitive theory and group dynamics, which will guide intrapersonal and interpersonal level intervention strategies. Integrated research-practice partnership models will guide strategies to address organizational and community-level influences.

The goal is to develop and test an adaptive randomized trial to enhance PA maintenance among cancer survivors. Our central hypothesis is that participants who have difficulty maintaining PA following a community-based exercise program will benefit from additional support in the form of bi-weekly exercise sessions and/or PA behavior change discussion sessions. Our long-term goal is to develop an evidence-based 'stepped' PA maintenance intervention for cancer survivors that can be disseminated to existing community-based cancer-exercise programs nationwide. In the proposed study, cancer survivors will participate in an existing, cancer-specific exercise program at a community-based facility.

All programs will consist of group-based, supervised, instructor-led aerobic and resistance exercise sessions 2x per week, and three PA behavior change discussion sessions. Upon completion of the program, participants will be encouraged to maintain PA levels during a three-month free-living period, during which time there will be no active intervention. After this follow-up period, PA will be measured, and based on PA response (i.e., achieving exercise guidelines for cancer survivors), participants will be randomized to a 3-month, stepped, PA maintenance intervention. The primary outcome of PA maintenance will be assessed six-months after completion of the initial exercise program.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old,
* Able to speak/read English,
* Diagnosed with any type of cancer,
* Completed primary or adjuvant treatment (i.e., chemotherapy, radiation therapy, surgery) within the previous five years, with no planned treatment within the next nine months. This does not include long-term or chronic therapies such as anti-hormone or targeted therapies (e.g., aromatase inhibitor, androgen deprivation therapy),
* Participant is registered/enrolled to participate in one of three community-based exercise programs.

Exclusion Criteria:

* Existing participation in ≥90 minutes per week of at least moderate intensity aerobic exercise AND two or more days per week of resistance exercise or known contraindications for exercise.
* Known contraindications for non-medically supervised moderate or greater intensity exercise (e.g., uncontrolled hypertension, inability to walk without an assistive device)
* Current or planned participation in another exercise oncology program (not one of the three community partner exercise programs), or previous participation in another or one of the three community partner exercise programs in the past 12-months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity program | Measured at baseline, after completion of the exercise program (either 8-weeks or 12-weeks), 3-months post program, and 6-months post program
  Examine the number of participants achieving the exercise guidelines for cancer survivors defined as moderate-intensity aerobic training at least three times per week, for at least 30 minutes, and resistance training at least two times per week. Aerobic exercise will be measured with an accelerometer (continuous bouts of ≥5 minutes of activity at ≥3 METs) and resistance exercise will be measured with a self-report questionnaire (duration and frequency). The measures will be aggregated to determine total amount of physical activity and whether this amount meets or exceeds the recommended guidelines.

SECONDARY OUTCOMES:
Quality of Life (QOL) | Measured at baseline, after completion of the exercise program (either 8-weeks or 12-weeks), 3-months post program, and 6-months post program
  Measured using the Functional Assessment of Cancer Therapy-General (FACT-G), a quantitative, self-report measure of QOL. The FACT-G is a 27-item self-report measure, with subscales evaluating physical, social, emotional, and functional well-being. FACT-G scores range from 0 to 108, with higher total and subscale scores indicating better QOL.
Physical Fitness - Aerobic | Measured at baseline, after completion of the exercise program (either 8-weeks or 12-weeks), 3-months post program, and 6-months post program
  Aerobic fitness will be assessed with either a submaximal, graded exercise test on a motorized, calibrated treadmill, or the two minute step test.
Physical Fitness - muscular strength and endurance | Measured at baseline, after completion of the exercise program (either 8-weeks or 12-weeks), 3-months post program, and 6-months post program
  Muscular strength and endurance will be assessed by the number of full stands from a chair, and the number of bicep curls (holding a hand weight of 5lbs) that can be completed in 30 seconds.

OTHER OUTCOMES:
Feasibility and acceptability of the PA maintenance intervention components | Through study completion, an average of 9-months
  Feasibility will include rate of recruitment, participant retention, completeness of data, and number of adverse events. Acceptability, among participants (i.e., cancer survivors) will be assessed via survey, and focus groups. Acceptability, implementation, and integration of the intervention among community facility leaders and fitness professionals will be assessed via semi-structured, face-to-face interviews which will focus on their satisfaction with the intervention delivery (i.e., cost, time, etc.), responses they observed from study participants, and sustainability within the organizational structure. Collectively, these outcomes will be aggregated to determine whether the maintenance intervention would be feasible to sustain in the community-based program.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Anschutz Medical Center, Aurora, Colorado
  - Colorado State University, Fort Collins, Colorado
  - University of Wyoming, Laramie, Wyoming

IPD SHARING:
Plan to Share IPD: No